CLINICAL TRIAL: NCT07211659
Title: A Phase I, Open-label, Dose Finding, Safety, Tolerability and Exploratory Trial of THEO-260 Administered Via an Intraperitoneal Route in Patients With High Grade Serous or Endometrioid Ovarian Cancer
Brief Title: Trial of THEO-260 (Administered Via Intraperitoneal Route) in Ovarian Cancer Patients
Acronym: OCTOPOD-IP
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Theolytics Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: THEO-260-002
Record Dates: First submitted 2025-10-01; First posted 2025-10-08 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Ovarian Cancer
Keywords: Ovarian cancer; Oncolytic virus; Intraperitoneal administration; Dose escalation
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- THEO-260 (Experimental)
  Interventions: Biological: THEO-260

INTERVENTIONS:
Biological: THEO-260 — Oncolytic virus

SUMMARY:
The goal of this clinical trial is to establish if THEO-260 is safe to administer to adult females with ovarian cancer. It will also aim to establish if THEO-260 is able to treat ovarian cancer. The main questions it aims to answer are:

* What medical problems do participants have when taking THEO-260?
* At what dose is THEO-260 both safe but also shows signs of being able to treat ovarian cancer?

The clinical trial follows a dose escalation/ finding design where we will aim to establish a Recommended Phase 2 Dose (RP2D).

Participants will:

* Be administered 6 doses of THEO-260 via an intraperitoneal (IP) route of administration over the course of 2 weeks.
* They will then visit the clinic at regular intervals for check-ups and tests to monitor safety and THEO-260 ability to treat ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed histological diagnosis of advanced high grade serous or endometrioid cancer of the fallopian tube, primary peritoneum or ovary either on archival biopsy or fresh tumour biopsy.
* Platinum-resistant or refractory disease: platinum-resistance is defined as radiological progression within 6 months of last cycle of platinum treatment; platinum refractory disease is defined as radiological progression during the 3 months following the first dose with platinum treatment.
* Voluntary, written informed consent prior to trial procedures. Willingness and ability to comply with the protocol.
* Life expectancy of > 6 months.
* Adequate haematological and organ function (parameters apply).
* Non-pregnant and non-lactating and surgically sterile, or post-menopausal or abstinent or if of child-bearing potential will to use a highly effective form of contraception - where applicable.
* ECOG performance status of 0 or 1.
* Measurable disease as per RECIST V1.1.

Exclusion Criteria:

* Prior anti-cancer treatment or receipt of investigational product within 28 days or 5 half-lives, prior to first dose of THEO-260 or patients with unresolved serious toxic side-effects of prior chemotherapy or radiotherapy.
* Prior treatment with a group B adenovirus.
* Currently enrolled in a clinical trial of an IP or used any IP with 5 half-live before screening.
* Radiation therapy within 4 weeks of first dose of THEO-260.
* Clinical evidence of cerebral metastases or Central Nervous System (CNS) involvement including leptomeningeal disease. Patients with previous cerebral metastases must have no evidence of progression or haemorrhage after treatment and have been off dexamethasone for 4 weeks prior to first dose of THEO-260 with no ongoing requirement for dexamethasone or anti-epileptic drugs. Brain imaging in patients with a history of cerebral metastases or CNS involvement must not be older than 12 weeks (at the start of screening). Results of any unexpected or abnormal findings of brain imaging should be discussed with the Medical Monitor and Sponsor as part of the screening process.
* Uncontrolled pleural effusion or pericardial effusion requiring recurrent drainage procedures (as defined as once monthly or more frequently).
* Prior pneumonitis or history of interstitial lung disease.
* Confirmed QTcF ≥470 ms on screening 12-lead ECG or history of Torsades de pointes or history of congenital long QT syndrome.
* Concomitant medications that prolong the QTc interval and/or increase the risk for Torsades de Pointes that cannot be discontinued or substituted (within 5 half-lives or 14 days prior to the first dose of IP, whichever was longer) with another drug prior to administration of IP.
* Any other concurrent severe and/or uncontrolled medical or surgical condition which, in the view of the Investigator, could compromise the patient's participation in the trial due to safety, compliance concerns or ability to evaluate response.
* Patients with active hepatitis infection (defined as having a positive hepatitis B surface antigen [HBsAg] test at screening) or hepatitis C.
* Active infection with tuberculosis. Past or resolved tuberculosis is acceptable.
* Active infection with severe acute respiratory syndrome coronavirus 2 (SARS-Cov-2). All patients should be tested for active SARS-Cov-2 infection and have a negative COVID-19 result within 3 days of Day 1 (e.g., if a patient tested positive in antigen testing but asymptomatic, the patient will need to be excluded). Active infection with SARS-Cov-2 confirmed as per site's standard way of testing.
* Patients with active human immunodeficiency virus (HIV) infection or known history of HIV infection.
* Active infection requiring IV antibiotics within 2 weeks prior to first dose of THEO-260, or long-term oral therapy for systemic infection.
* Known contra-indications or hypersensitivity to the excipients of the IP.
* Patients with an active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids, or immunosuppressive drugs).
* Known heart failure New York Heart Association (NYHA) Class 2-4.
* Any major surgical procedure (planned or anticipated) (in the Investigator's judgement) within 4 weeks of the first dose of THEO-260 or within the anticipated treatment period.
* Known contra-indications or hypersensitivity to acetaminophen.
* Known alcohol consumption in excess of 2 units per day.
* Patients with a left ventricular ejection fraction (LVEF) <45%, unstable angina, serious uncontrolled cardiac arrhythmia, a myocardial infarction within 6 months prior to trial enrolment or a history of myocarditis.
* Patients with arterial oxygen saturation <92% on room air prior to first dose of investigational product.
* Patients who have received any live vaccines within 30 days prior to enrolment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 18 (Estimated)
Dates: Start 2026-02-28 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of THEO-260 | Until end of trial for a participant, estimated at 1 year
  Safety and tolerability will be assessed by:
  Evaluation of DLTs and AEs during treatment and follow-up using National Cancer Institute (NCI) Common Terminology Criteria for AEs (CTCAE) v5.0 or American Society of Clinical Oncology (ASCO; for pneumonitis only) or American Society for Transplantation and Cellular Therapy (ASTCT; for cytokine release syndrome [CRS] only).
Establish recommended Phase 2 dose (RP2D) for THEO-260 | Until end of trial, estimated at 16 months after start of enrolment
  The totality of safety and efficacy data collected will be used to assess RP2D.

SECONDARY OUTCOMES:
Pharmacokinetic (PK) profile of THEO-260 | Until Day 29 after first dose
  Assess PK profile (maximum concentration - Cmax) of THEO-260 in blood by qPCR.
Shedding of THEO-260 in saliva, urine, and faeces | Until Day 29 after first dose
  Assess shedding of THEO-260 in buccal, urine and faecal samples by qPCR.
Risk of systemic cytokine release syndrome (CRS) after THEO-260 | Until Day 29 after first dose
  Assess systemic CRS following administration of THEO-260 by measurement of key markers in blood.
Evaluate preliminary efficacy of THEO-260 - RECIST | Until end of trial, estimated at 15 months after start of enrolment
  Determine response to THEO-260 as assessed by tumour imaging according to RECIST v1.1/iRECIST.
Evaluate preliminary efficacy of THEO-260 - CA125 | Until end of trial, estimated at 16 months after start of enrolment
  Efficacy will also be measured by changes in cancer antigen 125 (CA-125).

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Theolytics Ltd
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No